CLINICAL TRIAL: NCT00085852
Title: Phase 1 Study of the Aeris Bronchoscopic Lung Volume Reduction (BLVR) System in Patients With Advanced Heterogeneous Emphysema
Brief Title: US 10 mL Bronchoscopic Lung Volume Reduction (BLVR) Phase 1 Emphysema Study - Initial Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Edward P Ingenito, MD, PhD, Medical Director & CSO, Aeris Therapeutics Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C04-001; IRB Protocol # 2003-P-002171
Record Dates: First submitted 2004-06-15; First posted 2004-06-17 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Pulmonary Emphysema
Keywords: emphysema; chronic obstructive pulmonary disease; lung volume reduction; bronchoscopic; bronchoscopy; bronchoscope
MeSH Terms: conditions — Pulmonary Emphysema; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): Treatment with BLVR
  Interventions: Biological: BLVR

INTERVENTIONS:
Biological: BLVR — 10 mL Hydrogel

SUMMARY:
The purpose of this study is to determine whether the Aeris Bronchoscopic Lung Volume Reduction (BLVR) System is safe in patients with advanced emphysema.

DETAILED DESCRIPTION:
Patients with emphysema currently have limited treatment choices. Many patients are treated with steroids and inhaled medications, which often provide little or no benefit. Recently, lung volume reduction surgery has become an accepted therapy for emphysema. Lung volume reduction surgery involves the removal of a diseased portion of the lung, which enables the remaining, healthier portions of the lung to function better. This procedure, although effective, is complicated and risky.

Aeris Therapeutics has developed the Aeris Bronchoscopic Lung Volume Reduction System for treatment of patients with advanced emphysema. The Aeris BLVR System is designed to reduce lung volume without surgery. Patients are treated under anesthesia using a bronchoscope to direct treatment to the most damaged areas of the lung. The treatment is expected to reduce lung volume by shrinking the diseased areas of the lung. The purpose of the current study is to find out whether the Aeris BLVR System is safe in patients with advanced emphysema. The risks associated with the treatment are expected to be similar to those associated with general anesthesia and bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced emphysema
* Limited exercise capacity and persistent symptoms despite medical therapy
* Age between 18 and 75
* No significant heart, kidney or liver disease
* Willingness and ability to tolerate bronchoscopy
* No prior Lung Volume Reduction Surgery or Lung Transplantation
* Screening test results indicating that the procedure is appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
SAEs - Safety | 1 year post treatment

SECONDARY OUTCOMES:
PFTs | 12 weeks post treatment
Dyspnea | 12 weeks post treatment
Exercise capacity | 12 weeks post treatment
QOL | 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: John J. Reilly, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Caritas St Elizabeth's Medical Center, Boston, Massachusetts

REFERENCES:
- [Background] Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. doi: 10.1164/rccm.200208-842OC. Epub 2002 Oct 11. PMID 12406835